CLINICAL TRIAL: NCT05733676
Title: Comparison of MI Paste Plus and Resin Infiltration in Improvement of White Spot Lesions Following Fixed Orthodontic Treatment: A Randomized Controlled Trial
Brief Title: Comparison of MI Paste Plus and Resin Infiltration in White Spot Lesions Following Orthodontic Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAlberta-Pro00126739
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: White Spot Lesions; Orthodontic Appliance Complication; Caries Arrested; Smooth Surface Caries
Keywords: White spot lesion; caries; arrested; orthodontic
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: The selected samples will be randomly allocated to two groups according to treatment received.
  Group I- Resin infiltration -Icon + etch, DMG, Germany.
  Group II- MI paste plus +etch , GC corporation, Germany, Europe,
Who Masked: Participant, Outcomes Assessor
Masking Description: Double, Participant and Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin Infiltration (Active Comparator): Resin infiltration of early intervention of caries lesion as a consequences of orthodontic treatment
  Interventions: Device: Resin infiltration; Device: Casein Phosphopeptide (CPP) - Amorphous Calcium Phosphate (ACP) - Fluoride
- Casein Phosphopeptide (CPP) - Amorphous Calcium Phosphate (ACP) - Fluoride (Active Comparator): Casein Phosphopeptide (CPP) - Amorphous Calcium Phosphate (ACP) - Fluoride early intervention of caries lesion as a consequences of orthodontic treatment
  Interventions: Device: Resin infiltration; Device: Casein Phosphopeptide (CPP) - Amorphous Calcium Phosphate (ACP) - Fluoride

INTERVENTIONS:
Device: Resin infiltration — Base line treatment of white spot lesions in smooth surface with Resin infiltration -Icon + etch, DMG, Germany.
Device: Casein Phosphopeptide (CPP) - Amorphous Calcium Phosphate (ACP) - Fluoride — Base line treatment of white spot lesions in smooth surface with MI paste plus + etch , GC corporation, Germany, Europe

SUMMARY:
Dental cavities are among the most frequent diseases that affect teeth, particularly in patients who are treated with braces due to the difficulty in maintaining good oral hygiene in the presence of the mouth appliances. The white spot lesion (WSL) is the first clinical sign of cavities that presents itself as a milky-white opacity when located on the front face of the tooth. The aim to manage these early lesions focuses on promoting natural remineralization and preventing further demineralization. Various materials have been introduced for management of WSLs including MI paste and MI paste combined with fluoride (MI paste plus). Recently, a new material called resin infiltration has been found to treat these lesions with high esthetic results and great performance. According to the few numbers of in-vivo studies investigating the effectiveness of remineralization products, the aim of the current study is to clinically compare the outcome of the resin-infiltration and etching + MI paste plus to stop and improve the appearance of the WSL on front teeth in patients after treatment with braces.

DETAILED DESCRIPTION:
White spot lesion (WSL) is the first clinical sign of enamel caries that presents itself as a milky-white opacity non-cavitated when located on smooth surfaces. These surfaces are rougher than sound enamel, and they can be arrested or progressed. WSLs are more commonly seen on the outer surface of teeth after orthodontics treatment. Causing unaesthetic appearance on the anterior teeth and increasing chance of dental caries progression.

Different interventions have been introduced to manage WSL as preventing demineralization and biofilm formation, and promoting remineralization with fluoride varnish, casein phosphopeptides-amorphous calcium phosphate (CPP-ACP)- a nano-complex derived from milk casein that significantly increases salivary calcium and phosphate levels9 .

The remineralization of enamel subsurface lesions by CPP-ACP has been demonstrated in several in vitro studies. The potential of CPP-ACP to prevent enamel demineralization and promote lesion remineralization has also been successfully demonstrated in human in situ models. In the presence of fluoride, CPP-ACP has been shown to promote the formation of fluorapatite-like minerals deep in the subsurface lesion. Clinical studies evaluating the effect of CPP-ACP/ACFP on WSLs after debonding report significant regression of WSL numbers, size, and activity in comparison to fluoride or substances without fluoride. Consequently, CPP-ACP has been incorporated into minimally invasive products for the remineralization of WSLs. Nevertheless, other studies state significant change showing improvements in WSLs with remineralization products but no superiority of CPP-ACP .

Multiple studies have tested the efficacy of CPP-ACP on post-orthodontic WSLs but only a limited number of prospective clinical studies have examined the effect of CPP-ACP and fluoride + etch on WSLs developed during orthodontic treatment. It is during therapy with fixed appliances that patients are most susceptible to forming WSLs and WSLs are most active. Recently, treatment with resin infiltration has been developed by the dentistry equipe at Charité University of Berlin, Germany and was first proposed to halt the interproximal early stage non-cavitated caries lesions. It represents a new concept in dentistry that offers valuable clinical applicability for clinicians and high acceptance by patients and is an alternative method to treat early caries lesions that are not expected to remineralize or arrest by non-invasive measures when the infiltration is performed with low-viscosity light-curing resins.

The refractive index (RI) of enamel lesions is effective in arresting and stabilizing the progress of WSLs. Paris et al noted that lesions infiltrated by resin infiltration took on the appearance of the surrounding sound enamel masking the whitish appearance by filling the lesion's body with resin, which results in a rise of the refractive index (RI) of the lesion from 1-1. to 1.42-1.44 with resin infiltration, which is closer to a healthy enamel (1.62-1.63). Thus, a restoration with enamel-like optical characteristics is obtained. This technique is considered micro-invasive and may bridge the gap between the non-invasive and minimally invasive treatment of WSLs, postponing the need for a restoration as long as possible.

According to few in-vivo studies investigating the effectiveness of remineralization products to address the appearance of WSLs after orthodontic treatment.

The aim of the current study is to assess clinically the change in the WSL appearance of the maxillary incisors in patients treated with resin-infiltration + etch compared with patients treated with CPP-ACFP plus +etch .

Hypothesis: No significant difference will be expected between CPP-ACFP +etch (MI paste plus + etch) and resin infiltration etch in terms of improving the WSL however, the esthetic outcome of resin infiltration + etch will be significantly greater compared to MI paste plus + etch.

Justification: Few studies have evaluated in vivo the WSL change satisfaction of resin infiltration compared to CPP-ACP and fluoride + etch after orthodontic treatment for more than a year for follow ups. In-vitro and in-vivo studies have shown a change in WSLs as a result of the topical use of these materials. However, further studies are needed to prove their role in calcium-based remineralization systems.

Objectives:

Determine the effect of resin infiltration and CPP-ACP in the caries process Determine the effect of resin infiltration and CPP-ACP in incisors aesthetics

Methods:

In this clinical randomized controlled trial study, sixty two subjects in the age range of 12-21 years having at least one post-orthodontic WSL on the upper or lower incisors will be randomly assigned to two groups of 31 samples in each. Participants will be recruited from patients who underwent labial fixed orthodontic treatment with (bracket properties), bonded with light-cured composite resin adhesive (Transbond XT, 3M Unitek, U.S.A) in the Department of Orthodontics, Dental School, University of Alberta. The study period will be from March 2023 and so on with prior approval from IRB (HERB). Informed consents will be obtained from parents/caregivers of the children after explaining the details of the treatment procedure in a designated format in regional and English languages.

Justification of the sample size :

Using results from Baffif et al. (2020), sample size is estimated based on the effect size demonstrated from ICON as compared at the 6 month level is a mean difference of 0.8 with a standard deviation of 1.3. Assuming power of 0.8 and alpha of 0.05, the required sample size is 31 per group.The selected samples will be randomly allocated to two groups according to treatment received.

Group I- Resin infiltration -Icon + etch, DMG, Germany, (n=31). Group II- MI paste plus +etch , GC corporation, Germany, Europe, (n=31). Before the application of topical agents on white spot lesions, oral prophylaxis will be carried out and the affected tooth to be treated will be cleaned with a rubber cup with prophylaxis paste (3M, Clinpro, United States of America) in both groups.

Information in regards to the length of orthodontic treatment, date of removal of orthodontic appliances, and oral hygiene status during treatment will be collected from the patients' charts. Patients will randomly receive an 8-week regimen of MI paste plus or resin infiltration. Patients will be followed up at 3,6, 12 and 18 months to evaluate change in appearance of the lesion of both treatments.

Plan for Data Analysis:

Remineralization will be assessed by the enamel decalcification index score (EDI) and International caries detection and assessment system (ICDAS) to evaluate the WSLs change after treatment with the two remineralizing agents. Furthermore, the satisfaction evaluation of the lesion will be assessed by a Visual Analog Scale (VAS) from 0 mm no change to 100 mm WSL completely changed/disappeared. The assessment will be done with photographs. Intraoral frontal views will be taken digitally. These photographs will be obtained at baseline (a few days after debonding to allow resolution of gingival inflammation that might mask WSLs), 3, 6,12 and 18 months after completion of orthodontic treatment. The patients will be asked to tilt up their head approximately 5-10 degrees to limit the flash reflection to the incisal third of the maxillary incisors. The optimal image will be selected among several photographs that will be taken at each time point. The first panel will consist of 3 dental experts (orthodontists and pediatric dentists) while the second panel will consist of three laypersons. Each examiner will perform the assessment independently.

Statistical analysis:

The collected data will be subjected to statistical analysis using SPSS version 22.0 (Armonk, NY, IBM Corp). Demographic variables will be analyzed using proportions. Independent sample 't' test will be used to compare the mean difference in esthetic appearance (VAS) and lesion.

Repeated Measures ANOVA will be used to determine the mean difference in VAS and EDI score, within study groups at various time intervals.

Expected results No significant difference will be expected between MI paste plus+etch and resin infiltration etch in terms of improving the WSL; however, the esthetic outcome of resin infiltration + etch will be significantly greater compared to MI paste plus + etch.

Study significance WSLs are prevalent lesions on the surface of teeth particularly, around the attached brackets, which lead to unaesthetic appearance of teeth after bracket removal and increase the chance of initiation of dental caries. Caries in the anterior teeth compromise the aesthetic enhancement achieved by orthodontic treatment. Thus, introducing a material that changes the WSL while providing the most similar appearance to the tooth enamel will be of great value.

Risks and Discomforts This technique has no risk or discomfort during the research, as both materials have been approved in Canada. Except that the application of CCP-ACP + fluoride may be difficult for some people as they need to use it at home. This material is contraindicated in patients with a proven or suspected milk protein allergy and/or with a sensitivity or allergy to benzoate preservatives. No side effects have been reported so far.

During the study visits, there may be an increased risk of COVID-19 exposure due to the added time spent within our health care facility and possible exposure to others. All AHS Infection Prevention and Control Practices in place during the pandemic (screening for COVID 19 symptoms prior to hospital entry, use of masks, hand sanitizer and physical distancing measure where possible) will also apply during these visits to reduce COVID- 19 risks.

There may be risks in this study that are currently not known. If the investigators find out anything new during the course of this research which may change participants' willingness to be in the study, the investigators will tell participants about these findings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in the age range of 12-21 years who had undergone fixed orthodontic appliance therapy for a duration of 12-36 months.
* Should have at least one white spot lesion on the labial surface of either maxillary or mandibular anterior teeth after debonding. Lesion visible with or without drying the lesion surface.
* Patients with mild to moderate plaque accumulation. Fair oral hygiene. With a simplified Oral Hygiene Index of no more than 1.3-3.0

Exclusion Criteria:

* Poor oral hygiene Simplified Oral Hygiene Index of 3.1-6.0 or more
* Patients with hypoplasia or any developmental defects on the buccal of upper or lower incisors
* Patients with any restorations on the buccal of upper or lower incisors
* Patients that have presented WSL on the buccal of upper or lower incisors before orthodontic treatment was initiated.
* Patients that have received any re-mineralizing agent other than regular toothpaste during the last three months
* Patient with allergy to milk or any of their products
* Patient with any medical / oral or mental condition
* Patients or legal guardians that does not speak or read English

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Remineralization as assessed by the Enamel Decalcification Index (EDI) score with values 0-3 in each of the four tooth surfaces | 3 years
  Enamel decalcification index (EDI) score with values 0-3 in each of the four facial zones including mesial, distal, gingival, and occlusal surfaces around the approximate location of the debonded bracket it will represent the decalcification level based on clinical visual assessment of the tooth. The values will be recorded at baseline, 3, 6, 12,18 months. Tooth surfaces completely covered by gingiva or bonding material will be excluded. International caries detection and assessment system (ICDAS) with values 0-6 will be assigned to each tooth surface around the orthodontic bracket.
Satisfaction evaluation of the white spot lesion (WSL) as assessed by a Visual Analog Scale (VAS) from 0 mm no change to 100 mm completely changed | 3 years
  Intraoral frontal views will be taken at, 3, 6,12 and 18 months after completion of orthodontic treatment. This digital photography will be calibrated following protocols to standardize magnification, shade, and color. The images will be cropped to include the 4 incisors. Two independent, blinded panels will rate the WSL change using a visual analog scale (VAS) from 0 mm no change to 100 mm completely changed. The order of the participants will be shuffled so the bias resulted from examiner bias will be eliminated. The median value of the VAS will be selected as the representation for the percentage of change.

CONTACTS AND LOCATIONS:
Overall Officials: Ida M Kornerup, DMD, MEd, Principal Investigator — University of Alberta
Locations (1):
- KAYE Edmonton Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teshome A, Muche A, Girma B. Prevalence of Dental Caries and Associated Factors in East Africa, 2000-2020: Systematic Review and Meta-Analysis. Front Public Health. 2021 Apr 29;9:645091. doi: 10.3389/fpubh.2021.645091. eCollection 2021. PMID 33996722
- [Result] Cochrane NJ, Saranathan S, Cai F, Cross KJ, Reynolds EC. Enamel subsurface lesion remineralisation with casein phosphopeptide stabilised solutions of calcium, phosphate and fluoride. Caries Res. 2008;42(2):88-97. doi: 10.1159/000113161. Epub 2008 Jan 15. PMID 18204252
- [Result] Iijima Y, Cai F, Shen P, Walker G, Reynolds C, Reynolds EC. Acid resistance of enamel subsurface lesions remineralized by a sugar-free chewing gum containing casein phosphopeptide-amorphous calcium phosphate. Caries Res. 2004 Nov-Dec;38(6):551-6. doi: 10.1159/000080585. PMID 15528910
- [Result] Cai F, Manton DJ, Shen P, Walker GD, Cross KJ, Yuan Y, Reynolds C, Reynolds EC. Effect of addition of citric acid and casein phosphopeptide-amorphous calcium phosphate to a sugar-free chewing gum on enamel remineralization in situ. Caries Res. 2007;41(5):377-83. doi: 10.1159/000104796. PMID 17713338
- [Result] Huang GJ, Roloff-Chiang B, Mills BE, Shalchi S, Spiekerman C, Korpak AM, Starrett JL, Greenlee GM, Drangsholt RJ, Matunas JC. Effectiveness of MI Paste Plus and PreviDent fluoride varnish for treatment of white spot lesions: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Jan;143(1):31-41. doi: 10.1016/j.ajodo.2012.09.007. PMID 23273358
- [Result] Rechmann P, Bekmezian S, Rechmann BMT, Chaffee BW, Featherstone JDB. MI Varnish and MI Paste Plus in a caries prevention and remineralization study: a randomized controlled trial. Clin Oral Investig. 2018 Jul;22(6):2229-2239. doi: 10.1007/s00784-017-2314-9. Epub 2018 Jan 4. PMID 29299732
- [Result] Kielbassa AM, Muller J, Gernhardt CR. Closing the gap between oral hygiene and minimally invasive dentistry: a review on the resin infiltration technique of incipient (proximal) enamel lesions. Quintessence Int. 2009 Sep;40(8):663-81. PMID 19639091
- [Result] Askar H, Schwendicke F, Lausch J, Meyer-Lueckel H, Paris S. Modified resin infiltration of non-, micro- and cavitated proximal caries lesions in vitro. J Dent. 2018 Jul;74:56-60. doi: 10.1016/j.jdent.2018.03.010. Epub 2018 May 16. PMID 29775637
- [Result] Mazur M, Westland S, Guerra F, Corridore D, Vichi M, Maruotti A, Nardi GM, Ottolenghi L. Objective and subjective aesthetic performance of icon(R) treatment for enamel hypomineralization lesions in young adolescents: A retrospective single center study. J Dent. 2018 Jan;68:104-108. doi: 10.1016/j.jdent.2017.11.001. Epub 2017 Nov 28. PMID 29104142
- [Result] Paris S, Meyer-Lueckel H. Inhibition of caries progression by resin infiltration in situ. Caries Res. 2010;44(1):47-54. doi: 10.1159/000275917. Epub 2010 Jan 16. PMID 20090328
- [Result] Chen M, Li JZ, Zuo QL, Liu C, Jiang H, Du MQ. Accelerated aging effects on color, microhardness and microstructure of ICON resin infiltration. Eur Rev Med Pharmacol Sci. 2019 Sep;23(18):7722-7731. doi: 10.26355/eurrev_201909_18981. PMID 31599398
- [Result] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Result] Maheswari SU, Raja J, Kumar A, Seelan RG. Caries management by risk assessment: A review on current strategies for caries prevention and management. J Pharm Bioallied Sci. 2015 Aug;7(Suppl 2):S320-4. doi: 10.4103/0975-7406.163436. PMID 26538870
- [Result] Richter AE, Arruda AO, Peters MC, Sohn W. Incidence of caries lesions among patients treated with comprehensive orthodontics. Am J Orthod Dentofacial Orthop. 2011 May;139(5):657-64. doi: 10.1016/j.ajodo.2009.06.037. PMID 21536209
- [Result] Cruz CL, Edelstein BL. Linking orthodontic treatment and caries management for high-risk adolescents. Am J Orthod Dentofacial Orthop. 2016 Apr;149(4):441-2. doi: 10.1016/j.ajodo.2015.12.007. No abstract available. PMID 27021443
- [Result] Hagg U, Kaveewatcharanont P, Samaranayake YH, Samaranayake LP. The effect of fixed orthodontic appliances on the oral carriage of Candida species and Enterobacteriaceae. Eur J Orthod. 2004 Dec;26(6):623-9. doi: 10.1093/ejo/26.6.623. PMID 15650072
- [Result] Choi YY, Lee DY, Kim YJ. Colorimetric evaluation of white spot lesions following external bleaching with fluoridation: An in-vitro study. Korean J Orthod. 2018 Nov;48(6):377-383. doi: 10.4041/kjod.2018.48.6.377. Epub 2018 Sep 14. PMID 30450330
- [Result] Brochner A, Christensen C, Kristensen B, Tranaeus S, Karlsson L, Sonnesen L, Twetman S. Treatment of post-orthodontic white spot lesions with casein phosphopeptide-stabilised amorphous calcium phosphate. Clin Oral Investig. 2011 Jun;15(3):369-73. doi: 10.1007/s00784-010-0401-2. Epub 2010 Apr 10. PMID 20383545
- [Result] Reynolds EC. Remineralization of enamel subsurface lesions by casein phosphopeptide-stabilized calcium phosphate solutions. J Dent Res. 1997 Sep;76(9):1587-95. doi: 10.1177/00220345970760091101. PMID 9294493
- [Result] Oshiro M, Yamaguchi K, Takamizawa T, Inage H, Watanabe T, Irokawa A, Ando S, Miyazaki M. Effect of CPP-ACP paste on tooth mineralization: an FE-SEM study. J Oral Sci. 2007 Jun;49(2):115-20. doi: 10.2334/josnusd.49.115. PMID 17634723
- [Result] Kumar VL, Itthagarun A, King NM. The effect of casein phosphopeptide-amorphous calcium phosphate on remineralization of artificial caries-like lesions: an in vitro study. Aust Dent J. 2008 Mar;53(1):34-40. doi: 10.1111/j.1834-7819.2007.00006.x. PMID 18304239
- [Result] Reynolds EC, Cai F, Shen P, Walker GD. Retention in plaque and remineralization of enamel lesions by various forms of calcium in a mouthrinse or sugar-free chewing gum. J Dent Res. 2003 Mar;82(3):206-11. doi: 10.1177/154405910308200311. PMID 12598550
- [Result] Reynolds EC, Cai F, Cochrane NJ, Shen P, Walker GD, Morgan MV, Reynolds C. Fluoride and casein phosphopeptide-amorphous calcium phosphate. J Dent Res. 2008 Apr;87(4):344-8. doi: 10.1177/154405910808700420. PMID 18362316
- [Result] Shen P, Cai F, Nowicki A, Vincent J, Reynolds EC. Remineralization of enamel subsurface lesions by sugar-free chewing gum containing casein phosphopeptide-amorphous calcium phosphate. J Dent Res. 2001 Dec;80(12):2066-70. doi: 10.1177/00220345010800120801. PMID 11808763
- [Result] Manton DJ, Walker GD, Cai F, Cochrane NJ, Shen P, Reynolds EC. Remineralization of enamel subsurface lesions in situ by the use of three commercially available sugar-free gums. Int J Paediatr Dent. 2008 Jul;18(4):284-90. doi: 10.1111/j.1365-263X.2008.00920.x. Epub 2008 Apr 23. PMID 18435723
- [Result] Cai F, Shen P, Morgan MV, Reynolds EC. Remineralization of enamel subsurface lesions in situ by sugar-free lozenges containing casein phosphopeptide-amorphous calcium phosphate. Aust Dent J. 2003 Dec;48(4):240-3. doi: 10.1111/j.1834-7819.2003.tb00037.x. PMID 14738126
- [Result] Cochrane NJ, Shen P, Byrne SJ, Walker GD, Adams GG, Yuan Y, Reynolds C, Hoffmann B, Dashper SG, Reynolds EC. Remineralisation by chewing sugar-free gums in a randomised, controlled in situ trial including dietary intake and gauze to promote plaque formation. Caries Res. 2012;46(2):147-55. doi: 10.1159/000337240. Epub 2012 Apr 5. PMID 22488208
- [Result] Akin M, Basciftci FA. Can white spot lesions be treated effectively? Angle Orthod. 2012 Sep;82(5):770-5. doi: 10.2319/090711.578.1. Epub 2012 Feb 23. PMID 22356705
- [Result] Andersson A, Skold-Larsson K, Hallgren A, Petersson LG, Twetman S. Effect of a dental cream containing amorphous cream phosphate complexes on white spot lesion regression assessed by laser fluorescence. Oral Health Prev Dent. 2007;5(3):229-33. PMID 17977295
- [Result] Bailey DL, Adams GG, Tsao CE, Hyslop A, Escobar K, Manton DJ, Reynolds EC, Morgan MV. Regression of post-orthodontic lesions by a remineralizing cream. J Dent Res. 2009 Dec;88(12):1148-53. doi: 10.1177/0022034509347168. Epub 2009 Nov 3. PMID 19887683
- [Result] Wang JX, Yan Y, Wang XJ. Clinical evaluation of remineralization potential of casein phosphopeptide amorphous calcium phosphate nanocomplexes for enamel decalcification in orthodontics. Chin Med J (Engl). 2012 Nov;125(22):4018-21. PMID 23158136
- [Result] Singh S, Singh SP, Goyal A, Utreja AK, Jena AK. Effects of various remineralizing agents on the outcome of post-orthodontic white spot lesions (WSLs): a clinical trial. Prog Orthod. 2016 Dec;17(1):25. doi: 10.1186/s40510-016-0138-9. Epub 2016 Aug 2. PMID 27480987
- [Result] Beerens MW, van der Veen MH, van Beek H, ten Cate JM. Effects of casein phosphopeptide amorphous calcium fluoride phosphate paste on white spot lesions and dental plaque after orthodontic treatment: a 3-month follow-up. Eur J Oral Sci. 2010 Dec;118(6):610-7. doi: 10.1111/j.1600-0722.2010.00780.x. PMID 21083623
- [Result] Sabokseir A, Golkari A, Sheiham A. Distinguishing between enamel fluorosis and other enamel defects in permanent teeth of children. PeerJ. 2016 Feb 25;4:e1745. doi: 10.7717/peerj.1745. eCollection 2016. PMID 26966672
- [Result] Paris S, Hopfenmuller W, Meyer-Lueckel H. Resin infiltration of caries lesions: an efficacy randomized trial. J Dent Res. 2010 Aug;89(8):823-6. doi: 10.1177/0022034510369289. Epub 2010 May 26. PMID 20505049
- [Result] Senestraro SV, Crowe JJ, Wang M, Vo A, Huang G, Ferracane J, Covell DA Jr. Minimally invasive resin infiltration of arrested white-spot lesions: a randomized clinical trial. J Am Dent Assoc. 2013 Sep;144(9):997-1005. doi: 10.14219/jada.archive.2013.0225. PMID 23989837
- [Result] Bagher SM, Hegazi FM, Finkelman M, Ramesh A, Gowharji N, Swee G, Felemban O, Loo CY. Radiographic Effectiveness of Resin Infiltration in Arresting Incipient Proximal Enamel Lesions in Primary Molars. Pediatr Dent. 2018 May 15;40(3):195-200. PMID 29793566
- [Result] Giray FE, Durhan MA, Haznedaroglu E, Durmus B, Kalyoncu IO, Tanboga I. Resin infiltration technique and fluoride varnish on white spot lesions in children: Preliminary findings of a randomized clinical trial. Niger J Clin Pract. 2018 Dec;21(12):1564-1569. doi: 10.4103/njcp.njcp_209_18. PMID 30560818
- See also: Mi Paste Plus — https://www.gcamerica.com/downloads/SDS_CA/2018/SDS_CA_MI%20Paste%20Plus2.pdf